CLINICAL TRIAL: NCT03238820
Title: Robotic Resection for Patients With Gastric Gastrointestinal Stromal Tumors: a Single-center Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JIANG Zhi-Wei (Other)
Responsible Party: Sponsor-Investigator, JIANG Zhi-Wei, Vice director of Research Institute of General Surgery, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BE2015687GIST
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Gastrointestinal Stromal Tumor of Stomach
Keywords: Gastrointestinal stromal tumors; Robot; manual suture
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Intervention Model Description: This is a single group, open study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The robot group (Experimental): Patients undergo robotic gastric gastrointestinal stromal tumors resection.
  Interventions: Procedure: Robotic gastric gastrointestinal stromal tumors resection

INTERVENTIONS:
Procedure: Robotic gastric gastrointestinal stromal tumors resection — Robotic gastric gastrointestinal stromal tumors resection

SUMMARY:
Patients with gastric gastrointestinal stromal tumors will receive robotic resection.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumors are the most common stromal tumors of the digestive tract. Approximately 60% of tumors develop in the stomach.Before, patients with gastric gastrointestinal stromal tumors would receive open or laparoscopic surgery. However, gastrointestinal stromal tumors located at special sites, such as cardia, were hardly treated. Recently, the robot was used to remove gastric gastrointestinal stromal tumors. In this study, the robot will be used to remove gastric gastrointestinal stromal tumors. Then, we will evaluate the effect of robotic gastric gastrointestinal stromal tumors resection.

ELIGIBILITY:
Inclusion Criteria:

1. Requirements of informed consent and assent of participant, parent or legal guardian as applicable.
2. Patients with gastric gastrointestinal stromal tumors scheduled for robotic resection and between the age of 18 and 80 years old without considering sex.
3. American Society of Anesthesiologists (ASA) physical status I-III.
4. Participants can follow the visit plan.

Exclusion Criteria:

1. Patients certified by a doctor that doesn't fit to participate in this study.
2. Patients with ischemic heart disease, cerebrovascular disease and peripheral vascular disease, or their cardiac function > II (NYHA) patients, patients received coronary artery bypass grafting (CABG) recently, and patients with severe hypertension (systolic pressure≥180mmHg or diastolic pressure≥110mmHg).
3. Patients with gastrointestinal stromal tumor with distant metastasis.
4. Patients with severe infection, respiratory dysfunction, coagulation disorders, severe liver and renal dysfunction (Child - Pugh≥ 10; creatinine clearance < 25 ml/min).
5. Patients with gastrointestinal operations and complicated abdominal operations.
6. Patients with severe malnutrition (albumin≤30g/L, weight loss in half a year>10%, Subjective Global Assessment (SGA) classification C, body mass index <18, Hb<70g/L).
7. Pregnancy and lactation women, or have a pregnancy plan within a month after the test of the subjects (also including male participants).
8. Patients participated other subjects 3 months before this subject.
9. Sponsors or researchers directly involved in the testing or their family members.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Complications | 1 month
  Intraoperative and postoperative complications

SECONDARY OUTCOMES:
Blood loss | 1 day
  Blood loss
Operative time | 1 day
  Operative time
Resection style | 1 day
  The wedge resection, gastrotomy, partial gastrectomy and total gastrectomy were selected based on tumor size and site.
Postoperative length of stay | 1 month
  Postoperative length of stay
Inflammation level | 1 month
  Inflammation level
Nutritional status | 6 months
  Nutritional status
Body composition | 6 months
  Body composition

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Wei JIANG, Ph.D., Principal Investigator — Jinling Hospital, Medical School of Nanjing University; Jian ZHAO, Ph.D., Study Director — Jinling Hospital, Medical School of Nanjing University
Locations (1):
- Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
The results and IPD might be considered to share in published articles.